CLINICAL TRIAL: NCT03636334
Title: Learning Implementation of Guideline-based Decision Support System for Hypertension Treatment (LIGHT): A Staged Cluster Randomized Trial
Brief Title: Learning Implementation of Guideline-based Decision Support System for Hypertension Treatment (LIGHT)
Acronym: LIGHT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2016-I2M-1-006-1
Record Dates: First submitted 2018-07-03; First posted 2018-08-17 (Actual); Last update posted 2021-04-15 (Actual); Status verified 2021-04

CONDITIONS: Hypertension
Keywords: Hypertension; Decision support system; Staged cluster randomized controlled trial
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Computer-based decision support system (Experimental): Computer-based decision support system for BP management, with appropriate training of local PHC doctors.
  Interventions: Behavioral: Computer-based decision support system
- Control (No Intervention): After site randomization, physicians at the control sites will manage their patients with hypertension by usual care.

INTERVENTIONS:
Behavioral: Computer-based decision support system — At intervention sites, physicians will receive training and support on use of the DSS, which will be installed on their local IT system. Individuals eligible for DSS at Intervention sites will be randomized or assigned to different drug sequence protocols for BP-lowering therapy using their current antihypertensive medications, co-morbidities, and intolerance to medications and according to the assignment plan in the Algorithm. If the protocol is not suitable for the patient because of new co-morbidities, medication intolerance or contraindication, the DSS will recommend switching to a new protocol.
  Arms: Computer-based decision support system

SUMMARY:
This trial aims to evaluate the effectiveness of a guideline-based decision support system for hypertension management by physicians at primary health care (PHC) centers in China in order to improve the delivery of appropriate treatment and blood pressure (BP) control for hypertensive individuals.

DETAILED DESCRIPTION:
The LIGHT trial aims to assess the effectiveness of decision support system (DSS) for hypertension treatment in cluster clinics. At each stage, the main randomization will occur at the PHC center level. During the first 3 months (baseline period), the physicians at all sites will use an electronic data collection system to collect information about the individuals who attend the clinic. After site randomization, physicians at control sites will continue to deliver usual care, and physicians at intervention sites will receive training and support on the use of the DSS. And the DSS will recommend antihypertensive medications according to the assigned protocol. All individuals will be asked to attend the clinic at least once every 3 months.

ELIGIBILITY:
Inclusion Criteria for Sites:

1. At least one drug available from each of the four classes of recommended antihypertensive drugs are provided at clinic:

   * A: Angiotensin-converting enzyme inhibitors (ACEI; e.g., captopril and nalapril) or angiotensin receptor blockers (ARB; e.g., losartan and valsartan)
   * B: β-blockers (e.g., atenolol and metoprolol)
   * C: Calcium antagonists (e.g., nitrendipine, nifedipine, and amlodipine)
   * D: Diuretics (e.g., hydrochlorothiazide and indapamide)
2. Has an outpatient clinic for hypertension treatment and staff willing to take part in the study
3. Electronic data collection system is routinely used at clinic for hypertension management
4. At least 100 individuals with hypertension can attend the clinic every 3 months.

Inclusion Criteria for Visits:

1. Scheduled or unscheduled visit for hypertension treatment or prescription for antihypertensive medications
2. Visit for elevated blood pressure or adverse effect of antihypertensive medications
3. Visit for other cardiovascular diseases such as diabetes, stroke, PAD, or newly diagnosed of CKD, CAD and heart failure regardless of individuals' blood pressure level.

Inclusion Criteria for Participants:

1. Age ≥18 years
2. Local resident of the community/township who attend the PHC clinic for hypertension management
3. Established diagnosis of essential hypertension (defined as systolic blood pressure≥140 mmHg, diastolic blood pressure ≥90 mmHg, or both, measured on at least 3 separate visits; or currently taking antihypertensive medications)
4. Taking 0-2 types of antihypertensive medications (not including B)

Exclusion Criteria for participants:

1. Patients with SBP≥180 mmHg and/or DBP≥110 mmHg
2. History of coronary heart disease (i.e., angina, MI, coronary artery bypass grafting [CABG], percutaneous coronary intervention [PCI], >50% stenosis of coronary artery, or positive stress test)
3. Physician- diagnosed heart failure
4. Physician-diagnosed or self-reported CKD, estimated glomerular filtration rate (eGFR) <60 mL/min/1.73 m2 (if serum creatinine is available), or currently on dialysis
5. Physician-diagnosed secondary hypertension
6. Intolerance to at least two classes of antihypertensive medications among A, C or D
7. Other serious medical illness such as malignant cancer, hepatic dysfunction, et al
8. Currently at the acute phase of any disease
9. Subject is pregnant or breast feeding, or planning to become pregnant or breast feeding during study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10000 (Estimated)
Dates: Start 2019-08-21 (Actual); Primary Completion 2022-03-30 (Estimated); Study Completion 2022-03-30 (Estimated)

PRIMARY OUTCOMES:
The proportion of visits with ideal appropriate treatment provided among all the eligible hypertension visits within the period of observational follow-up | Baseline; 1 year
  ideal appropriate treatment means guideline-accordant treatment

SECONDARY OUTCOMES:
The average change in SBP from first visit after randomization to the last visit among the eligible participants during the period of 9-month observation. | Baseline; 1 year
  the average change in SBP from first visit after randomization to the last visit among enrolled patients.
The percentage of participants with BP<140/90 mmHg at the last visit among the eligible participants during the period of 9-month observation. | Baseline; 1 year
  The individuals' last blood pressure measurement during the 9-month observation phase will be used for assessment
The proportion of visits with acceptable appropriate treatment among all the eligible hypertension visits. | Baseline; 1 year
  Acceptable appropriate treatments is defined as the recommendations offered by the doctors who are not following DSS on reasonable conditions, such as patient-reported normal home-measured blood pressure, hypotension or syncope before the visit.

OTHER OUTCOMES:
The proportion of individuals with a vascular event (defined as cardiac death, non-fatal stroke and non-fatal MI) at 1 year. | Baseline; 1 year
  Measure the proportion of individuals who complicate with a vascular event.

CONTACTS AND LOCATIONS:
Overall Officials: Xin Zheng, MD, PhD, Principal Investigator — National Center for Cardiovascular Diseases
Locations (3):
- China (3):
  - Luoyang Oriental hospital, Beijing, Henan
  - Yankuang Hospital, Zoucheng, Shandong
  - Center for chronic disease control, Shenzhen, Shenzhen

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Song J, Wang X, Wang B, Ge Y, Bi L, Jing F, Jin H, Li T, Gu B, Wang L, Hao J, Zhao Y, Liu J, Zhang H, Li X, Li J, Ma W, Wang J, Normand ST, Herrin J, Armitage J, Krumholz HM, Zheng X; LIGHT Collaborative Group. Learning implementation of a guideline based decision support system to improve hypertension treatment in primary care in China: pragmatic cluster randomised controlled trial. BMJ. 2024 Jul 23;386:e079143. doi: 10.1136/bmj-2023-079143. PMID 39043397
- [Derived] Yi J, Wang L, Song J, Liu Y, Liu J, Zhang H, Lu J, Zheng X. Development of a machine learning-based model for predicting individual responses to antihypertensive treatments. Nutr Metab Cardiovasc Dis. 2024 Jul;34(7):1660-1669. doi: 10.1016/j.numecd.2024.02.014. Epub 2024 Mar 4. PMID 38555240
- [Derived] Song J, Wang X, Wang B, Gao Y, Liu J, Zhang H, Li X, Li J, Wang JG, Cai J, Herrin J, Armitage J, Krumholz HM, Zheng X; LIGHT Collaborative Group. Effectiveness of a clinical decision support system for hypertension management in primary care: study protocol for a pragmatic cluster-randomized controlled trial. Trials. 2022 May 16;23(1):412. doi: 10.1186/s13063-022-06374-x. PMID 35578345